CLINICAL TRIAL: NCT05231681
Title: Study to Identify if Saie Beauty's Under Eye Concealer Works to Improve Under-Eye Skin Appearance and Reduce Imperfections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saie Beauty (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20231Saie
Record Dates: First submitted 2022-01-31; First posted 2022-02-09 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Wrinkle
Keywords: skin aging; fine lines; crow's feet; dark circles

STUDY DESIGN:
Intervention Model Description: This is an open-label single-group, non-randomized, non-controlled interventional treatment study.
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eye Concealer (Experimental): Saie Beauty's Hydrabeam Sheer Brightening Under Eye Concealer
  Interventions: Dietary Supplement: Saie Beauty's Hydrabeam Sheer Brightening Under Eye Concealer

INTERVENTIONS:
Dietary Supplement: Saie Beauty's Hydrabeam Sheer Brightening Under Eye Concealer — Eye Concealer

SUMMARY:
Saie Beauty has developed 'Hydrabeam Sheer Brightening Under Eye Concealer' that is specifically designed for improving under-eye skin health. The concealer is aimed at improving under-eye skin features including hydration, firmness/elasticity, smoothness, and brightness. At the same time, it is aimed at reducing imperfections such as dark circles, skin redness, fine lines, wrinkles, and crow's feet. The aim is to understand and assess the efficacy of treatment from the participants' perspective and to see if the participants reported changes in skin features, dark circles, brightness, fine lines, wrinkles, crow's feet, and other skin imperfections.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 45 years old
* Must be in good general health
* Want to improve under-eye skin health by improving skin hydration, firmness/elasticity, smoothness, and brightness
* May have dark circles, fine lines, wrinkles, and crow's feet
* Must be willing to comply with the study protocol
* Must be willing to add the concealer to their daily routine for the duration of the study
* Must maintain a basic skincare routine, e.g., must use moisturizer and sunscreen daily
* Able to communicate in English
* Must provide a written Informed Consent Form (ICF)
* Willing to share feedback via the given online portal

Exclusion Criteria:

* Unwilling to follow the routine of the study
* Unwilling to provide informed consent
* Currently participating in another research study
* Severe chronic conditions including ontological and psychiatric conditions
* Use of prescription medication relevant for the skin
* Have any known allergies to the ingredients of the test product
* Known to have any severe allergic reactions in the past
* Undergoing any cosmetic procedures such as laser treatments, Botox, or chemical peels for the duration of the study.
* Have diagnosed or self-identified sensitive skin
* Have any learning and/or cognitive difficulties that prevent them from reading and understanding questionnaires and surveys (e.g. dementia)
* Currently pregnant or breastfeeding, or want to become pregnant for the duration of the study
* Use of prescription drugs (topical or oral) that are targeted at any sort of skin condition (for example retinoids)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Based on gender identity
Enrollment: 35 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Skin aging [Time frame: Baseline to 4 weeks] | 4 weeks
  Patient reported outcome measures (Scale 0-5 with higher scores representing a better outcome) to assess the reduction of early signs of aging such as fine lines, dark spots, and brighter skin

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Mitschke, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided